CLINICAL TRIAL: NCT00904904
Title: Indomethacin Eyedrops Compared With Ketorolac Eyedrops for Ocular Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 539; 2007-004686-18 (EudraCT Number)
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Cataract; Inflammation
MeSH Terms: conditions — Cataract; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indomethacin (Experimental): Indomethacin ophthalmic solution 0.1% for post-surgical inflammation
  Interventions: Drug: Indomethacin ophthalmic solution
- Ketorolac (Active Comparator): Ketorolac ophthalmic solution 0.5% for post-surgical inflammation
  Interventions: Drug: Ketorolac Ophthalmic Solution

INTERVENTIONS:
Drug: Indomethacin ophthalmic solution — Indomethacin 0.1% eye drops administered pre-cataract surgery and for 4 weeks post-cataract surgery
  Arms: Indomethacin
Drug: Ketorolac Ophthalmic Solution — Ketorolac 0.5% eye drops administered pre-cataract surgery and 4 weeks post-cataract surgery
  Arms: Ketorolac

SUMMARY:
This study is being conducted to show that indomethacin is at least as effective as ketorolac for the prevention of ocular inflammation following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be planning to undergo cataract surgery on one eye by phacoemulsification with posterior chamber intraocular lens, using topical or general anaesthesia.
* Subjects must have a preoperative flare ≤ 15 ph/ms, measured with a laser flare meter(LFM) without pharmacological pupil dilation, within the 2 months preoperatively.

Exclusion Criteria:

* Subjects who have any progressive pathology requiring the use of topical or systemic anti-inflammatory or anti-infectious agents.
* Subjects who take acetylsalicylic acid at doses > 100 mg daily and cannot discontinue usage during the study.
* Subjects who have a history of asthma linked to acetylsalicylic acid or other nonsteroidal anti-inflammatory (NSAI) drug administration.
* Subjects with immunodepression.
* Subjects with a history of intolerance to the study drug or to any NSAI drug.
* Subjects who are monocular for any reason other than cataract.
* Subjects who are treated with local or systemic anti-inflammatory drugs within 10 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Aqueous flare | Post-operative day 1 & day 7

SECONDARY OUTCOMES:
Aqueous flare | Postoperative day 30 and day 90
Change from baseline of retinal thickness | Postoperative day 30 & day 90

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Brenger, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Berlin, Germany